CLINICAL TRIAL: NCT01502995
Title: Laser Light Visual Cueing for Freezing of Gait in Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Parkinson's Disease Research, Education, and Clinical Center, Philadelphia (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 00583
Record Dates: First submitted 2011-12-21; First posted 2012-01-02 (Estimated); Last update posted 2012-01-02 (Estimated); Status verified 2011-12

CONDITIONS: Parkinson Disease
Keywords: Assistive devices; Freezing of gait; Gait disorders; Gait hesitation; Gait ignition failure; Laser light; Parkinson's disease; Rolling walker; Visual Cue; Walker
MeSH Terms: conditions — Parkinson Disease; Mobility Limitation | interventions — Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- With laser light (Active Comparator): Trial of walking tasks using laser light on walker.
  Interventions: Device: Laser light (U-Step Walking Stabilizer with laser light)
- Without laser light (Active Comparator): Trial of walking task without laser light on walker.
  Interventions: Device: Laser light (U-Step Walking Stabilizer with laser light)

INTERVENTIONS:
Device: Laser light (U-Step Walking Stabilizer with laser light) — Use of a laser light on a rolling walker during episodes of freezing of gait.
  Other Names: U-Step Walking Stabilizer with laser light

SUMMARY:
The purpose of this study is to determine whether a laser light beam, attached to a rolling walker and projected onto the floor, reduces freezing episodes in patients with Parkinson's disease.

DETAILED DESCRIPTION:
Freezing of gait is a debilitating feature of Parkinson's disease. This study aims to determine whether a laser light beam, attached to a rolling walker and projected onto the floor, reduces freezing episodes. Patients will perform two trials of 3 timed walking tasks: once with the laser beam and once without. For each trial, the time to complete, number of steps, and number of freezing episodes will be recorded. Patients will be randomized to perform the first trial either with the light or without the light, to control for fatigue.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic PD confirmed by a movement disorders neurologist
* a Mini-Mental Status Examination (MMSE)[13] score ≥ 24 to ensure competence to participate in informed consent and an ability to learn procedurally the use of the rolling walker with laser beam
* functional visual acuity for recognizing the laser beam on the rolling walker
* FOG in both on and off medication states, as indicated by a score of ≥ 2 on Item 14 of the Unified Parkinson's Disease Rating Scale (UPDRS) and/or ≥1 on Item 3 of the Freezing of Gait Questionnaire (FOGQ)
* ability to ambulate for at least household distances with or without an assistive device as indicated by scoring 0, 1, or 2 on Items 15 and 29 of the UPDRS.

Exclusion Criteria:

* diagnosis of a gait disorder other than Parkinson's disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2003-06; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Time to complete walking task | Two hours
  Time in seconds for subject to complete the designated walking task.

SECONDARY OUTCOMES:
Number of steps | Two hours
  Number of steps taken to complete the designated walking task.
Number of freezing episodes | Two hours
  Number of freezing episodes that occur during walking task.

CONTACTS AND LOCATIONS:
Overall Officials: Lisette Bunting-Perry, PhD, RN, Principal Investigator — Philadelphia VAMC PADRECC
Locations (1):
- Philadelphia VA Medical Center PADRECC, Philadelphia, Pennsylvania, United States